CLINICAL TRIAL: NCT06762717
Title: Real World Data Collection in Chinese Population Treated With the FARAPULSE™ Pulsed Field Ablation System
Brief Title: FARAPULSE™ Pulsed Field Ablation System
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF333
Record Dates: First submitted 2025-01-06; First posted 2025-01-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: FARAPULSE™ Pulsed Field Ablation system — no intervention design in the study

SUMMARY:
To obtain real world data on the use of, and provide continued evidence on safety and effectiveness of the FARAPULSE™ Pulsed Field Ablation (PFA) system when used per hospitals' standard of care in Chinese population.

DETAILED DESCRIPTION:
The study is an observational, prospective, non-randomized, single-arm, multi-center post-market study.

All subjects signing the informed consent form, will be included in the study. All subjects treated with the FARAPULSE™ PFA system will be followed for three years.

Subjects will undergo the index procedure per hospitals' standard of care after enrollment, and followed at pre-discharge, 3 Month, 6 Month (Phone call only), 12 Month (in-clinic visit mandatory), 24 Month (2 Year) and 36 Month (3 Year).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects intended to be treated with the FARAPULSE™ Pulsed Field Ablation system for cardiac tissue ablation, per physician's medical judgement, and as per hospitals' standard of care
2. Subjects who are willing and capable of providing informed consent
3. Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center
4. Subjects whose age is 18 years or above.

Exclusion Criteria:

1. Subjects with a current interatrial baffle or patch
2. Subjects with a known or suspected atrial myxoma
3. Subjects with a myocardial infarction within 14 days prior to enrollment
4. Subjects with a recent (within 30 days prior to enrollment) Cerebral Vascular Accident (CVA)
5. Subjects who do not tolerate anticoagulation therapy
6. Subjects with an active systemic infection *
7. Subjects with a presence of atrial known thrombus *
8. Subjects with a known inability to obtain vascular access
9. Subjects who are pregnant or planning to be pregnant
10. Subjects with atrial fibrillation that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
11. Subjects with any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty
12. Subjects with a contraindication to an invasive electrophysiology procedure where insertion or manipulation of a catheter in the cardiac chambers is deemed unsafe per physician's medical judgement, such as, but not limited to, a recent previous cardiac surgery (e.g., ventriculotomy or atriotomy, CABG, PTCA/PCI/coronary stent procedure), recent previous unstable angina and/or in patients with congenital heart disease where the underlying abnormality increases the risk of the ablation (e.g., severe rotational anomalies of the heart or great vessels)
13. Subjects with a life expectancy of ≤ 1 year per investigator's opinion
14. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the FARADISE study will be clinically indicated for an ablation procedure with the FARAPULSE™ Pulsed Field Ablation system, per indication approved in China, per physician's medical judgement, and according to hospitals' standard of care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure-free rate | 12 Months
  Failure-free rate at 12 Month post index procedure.
Device-or procedure-related SAEs: | 7 days and 12 months
  Composite of the following device- or procedure-related SAEs:
Procedure- and device related adverse events | 12 Months and 2 years and 3 years
  All FARAPULSE™ PFA procedure- and device related adverse events at 12 Month, 2 Year and 3 Year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Min Tang, Dr, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China/Beijing, China